CLINICAL TRIAL: NCT01579344
Title: Lacrimal Drainage System Obstruction Associated to Radioactive Iodine Therapy for Thyroid Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fabricio Lopes da Fonseca (Other)
Responsible Party: Sponsor-Investigator, Fabricio Lopes da Fonseca, Principal Investigator, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0528/11
Record Dates: First submitted 2012-04-15; First posted 2012-04-17 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Lacrimal Apparatus Disease
Keywords: Iodine Radioisotopes; Nasolacrimal Duct; radiation effects
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thyroid carcinoma, Radioactive iodine therapy (Active Comparator): 50 patients (100 eyes) diagnosed with differentiated thyroid carcinoma undergoing radioactive iodine therapy
  Interventions: Drug: Radioiodine therapy
- Thyroid carcinoma, without radioactive iodine therapy (No Intervention): 50 patients (100 eyes) diagnosed with differentiated thyroid carcinoma not undergone radioactive iodine therapy

INTERVENTIONS:
Drug: Radioiodine therapy — Radioiodine therapy with NaI131
  Arms: Thyroid carcinoma, Radioactive iodine therapy

SUMMARY:
The radioactive radioiodine therapy (Na131I) for the treatment of differentiated thyroid carcinoma is a procedure used for ablation of remaining thyroid tissue after thyroidectomy and metastases. Although serious complications are uncommon after treatment, there are well-documented adverse reactions secondary to the involvement of the salivary glands, such as dry mouth, pain in the parotid glands and dysphagia, even after administration of low doses of radioiodine. However, ocular complications of such treatment are scarcely reported in literature.

Among them the investigators can mention recurrent and chronic conjunctivitis, keratoconjunctivitis sicca and dry eye, affecting 23% of patients undergoing radioactive iodine therapy. Dysfunction of the lacrimal gland is described in recent studies, especially after high cumulative dose of the drug. Likewise, epiphora and nasolacrimal duct obstruction have been reported as complications associated with the use of radioiodine, although studies are not available to assess its true incidence through the systematic evaluation of patients.

It can be seen in routine practice that these patients would normally be referred for ophthalmological examination only if a complaint, what happens in the process of OVL already installed after the use of high doses of radioiodine. With the early evaluation of these patients, the investigators focused on detecting the process of ongoing obstruction in order to study interventions that prevent its final installation.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid carcinoma
* Previous thyroidectomy

Exclusion Criteria:

* Potential causes of dry eye (autoimmune diseases, contact lens wearers or drugs that alter tear production, such as antihistamines and psychotropic)
* Use of other anti-neoplastic, such as 5-fluorouracil and docetaxel, which can cause epiphora and OVL
* Lacrimal gland / ocular trauma
* Radiation therapy for other diseases or radiotherapy of head and neck
* Patients with diseases that alter the neural control of tear secretion, hormone therapies, pterygium, Graves' disease with or without ophthalmopathy, blepharitis and other conditions that may reduce tear production or result in rapid evaporation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Suzana Matayoshi, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo; Ophthalmology Department, São Paulo, São Paulo, Brazil